CLINICAL TRIAL: NCT04473495
Title: The Impact of Video Information on Preoperative Anxiety in Interventional Cardiology Patients.
Acronym: VATIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI013
Record Dates: First submitted 2020-05-05; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- video: patients who enjoyed an educational video
  Interventions: Device: educational video
- control: patients who didn't enjoy any educational video

INTERVENTIONS:
Device: educational video — educational video before intervention
  Groups: video

SUMMARY:
This study evaluates the impact of educative videos on anxiety for patients entering hospital for cardiology intervention

ELIGIBILITY:
Inclusion Criteria:

* patient entering hospitalisation in cardiology department for a cardiology intervention.

Exclusion Criteria:

* protected person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient entering hospitalisation in cardiology department for a cardiology intervention
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
anxiety | 1 year
  anxiety measured with STAI Y-A questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Sellal, Principal Investigator — Central Hospital, Nancy, France